CLINICAL TRIAL: NCT00946582
Title: The Therapeutic Effects of Barkley's Parenting Management Program for Taiwanese School-aged Children With Attention Deficit/Hyperactivity Disorder
Brief Title: The Therapeutic Effects of Barkley's Parenting Management Program for Taiwanese School-Aged Children With Attention Deficit/Hyperactivity Disorder (ADHD)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Liu, Shu-Tsen, Department of Psychiatry, National Taiwan University Hospital, Yun-Lin Branch
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200904005R
Record Dates: First submitted 2009-07-23; First posted 2009-07-27 (Estimated); Last update posted 2009-07-27 (Estimated); Status verified 2009-07

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: parenting management program; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Barkley's parenting management program — It is a parent training group to teach behavior therapy techniques to parents of children with ADHD. The group will contain about 10 parents of children with ADHD. It will be conducted 1.5 hour per session, one session per week, and 11 sessions totally.

SUMMARY:
The purpose of this study is to explore the therapeutic effects of Barkley's parenting management program for Taiwanese school-aged children with ADHD. The investigators hypothesized that Barkley's parenting management program might empower the parents' competence to manage their school-aged children's ADHD-related disturbing behaviors as its previously-proven effects for parents and their preschool-aged children with ADHD.

DETAILED DESCRIPTION:
Participants will be recruited from the child psychiatric clinics of NTUH-Yunlin branch and will include 30 school children with ADHD, their parents and teachers. The Kiddie-Schedule for Affective Disorders and Schizophrenia-epidemiology version will be adopted to confirm the diagnosis of ADHD. The child participants will received assessments of the Conner's Continuous Performance Test, and the Wechsler Intelligence Scale for Children-4th edition. We use ADHD symptoms, children't wellbeing, parent-child relationship, parent's competence and parenting stress as the outcome indices of therapeutic effects.Research instruments employed include CBCL, SNAP-IV, Parental Bonding Instrument, The Family Adaptability and Cohesion Evaluation Scale, Chinese Health Questionnaire, Parenting Stress Index, Short Form, Multidimensional student's life satisfaction scale and Nowicki-Strickland Locus of Control Scale for Children.

ELIGIBILITY:
Inclusion Criteria:

* Parents of 7-12 year-old aged children with ADHD and overall normal intelligence

Exclusion Criteria:

* Parents of children with comorbid autism spectrum disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
SNAP-IV | pretest, before session 4, before session 8, posttest, 3 months after the program finished

SECONDARY OUTCOMES:
Parenting Stress Index, Short Form | pretest, posttest, 3 months after the program finished

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Tsen Liu, M.D, Study Director — Department of Psychiatry, National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital Yun-Lin Branch, Douliu, Yunlin County, Taiwan